CLINICAL TRIAL: NCT02211105
Title: Laparoscopic Nissen Fundoplication (LNF) Surgery Versus Transoral Incisionless Fundoplication (TIF): Anti- Reflux Treatment Registry
Brief Title: Registry to Compare Two Surgical Treatments for GERD
Acronym: STAR Registry
Status: Terminated | Type: Observational
Why Stopped: Unexpected low accrual
Sponsor: American Gastroenterological Association (Other)
Collaborators: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA STAR Registry
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-04

CONDITIONS: GastroEsophageal Reflux Disease
Keywords: GastroEsophageal Reflux Disease; Transoral Incisionless Fundoplication; Laparoscopic Nissen Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laparoscopic Nissen Fundoplication: Patients whose GERD is being treated surgically through Laparoscopic Nissen Fundoplication.
- Transoral Incisionless Fundoplication: Patients whose GERD is being treated surgically through Transoral Incisionless Fundoplication.

SUMMARY:
The purpose of this prospective observational research study registry is to examine whether two GERD surgeries (Laparoscopic Nissen Fundoplication (LNF) or Transoral Incisionless Fundoplication (TIF)) have similar outcomes in effectiveness, safety, post-operative side effects and post-procedure costs associated with episodes of care and any ensuing complications.

DETAILED DESCRIPTION:
This registry will prospectively enroll 500 patients undergoing TIF and LNF from approximately 20 United States centers proficient in these procedures that have provided informed consent for the above mentioned data collection (symptom questionnaires, medical treatments, complications, side-effects and costs). The observational registry will obtain the patients clinical data related to gastrointestinal symptoms for three years post-consent.

At baseline and for a three-year period following a clinically indicated TIF or LNF procedure, data will be obtained from phone calls and/or during office-visits made at specified intervals. During these data collection periods, patients will be asked to complete standard validated symptom questionnaires as well as report on episodes of care related to their procedures along with financial costs of care.

ELIGIBILITY:
Inclusion Criteria:

* GERD symptoms (heartburn, defined by a sub-sternal burning discomfort arising from the upper abdomen into the chest, and or regurgitation, defined as the effortless arising of liquid material into the chest or mouth) two or more times a week (when not on anti-secretory medication) that adversely affects the patient's quality of life. Additionally, patients will have to have responded to medical therapy (adequate relief of symptoms) as indicated by GERD-HRQL and regurgitation scores on medical therapy. In this context, scores ≤ 2 on each GERD-HRQL and regurgitation question (while on medication) indicate absence of daily bothersome symptoms and therefore these patients are considered responsive to medical therapy. Furthermore, patients will have to have objective evidence of GERD documented (esophagitis on endoscopy or pathological intraesophageal acid exposure on prolonged ambulatory esophageal pH monitoring).
* Age 18-80 years
* Ability to give informed consent
* Regular access to a telephone
* Meet the clinical criteria for treatment of GERD with TIF or LNF and undergo TIF or LNF within 90 days of providing consent.

  * Dependent upon PPIs for control of heartburn for > six months or patient determined to have an inadequate response of regurgitation symptoms despite heartburn control with PPIs
  * Hiatal hernia axial length is no larger than 2 cm and the transverse dimension should not exceed 2.0 cm
  * Gastroesophageal junction with a Hill Grade I-II

    --- Patient willing to provide informed consent, cooperate with post-operative dietary recommendations and follow-up assessment tests
  * Objective documentation of pathological acid-reflux by either a) increased intraesophageal acid exposure on prolonged ambulatory esophageal pH monitoring (pH<4 for 4.5% or greater of the time) with or without impedance b) or the presence of erosive esophagitis (LA Grade A or B) on endoscopy
  * Absence of a severe esophageal motility disorder (note: mild abnormalities in esophageal motility are common in GERD such as small breaks, etc.) including achalasia, esophagogastric junction outflow obstruction, frequent failed peristalsis, diffuse esophageal spasm, nutcracker or jackhammer esophagus etc. on high-resolution esophageal manometry using the Chicago classification system or evidence of incomplete bolus clearance on 30% or more of swallows by impedance testing.

Exclusion Criteria:

* Hiatal hernia > 2 cm (defined as longitudinal length measured endoscopically between the proximal margin of the gastric folds and the diaphragmatic pinch)
* Esophagitis LA Grade C or D
* Presence of troublesome atypical symptoms
* Barrett's esophagus greater than 2 cm in length or with any dysplasia
* Esophageal stricture or severe esophageal motility disorder
* History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, cirrhosis or any other uncontrolled systemic disease

  --. Active gastro-duodenal ulcer disease
* Gastric outlet obstruction or stenosis
* Gastroparesis or delayed gastric emptying confirmed by a four hour solid-phase gastric emptying study
* Body Mass Index (BMI) > 35
* Pregnancy or plans for pregnancy within 12 months of the procedure
* Portal hypertension and/or varices
* New York Heart Association classification of III or IV.
* Coagulation disorders
* Intraprocedural determination of anatomical presentation which in the opinion of the surgeon does not allow safe performance of the procedure
* Enrollment in another device or drug study that may confound result

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who meet clinical criteria and have decided to treat their GERD through one of two surgical procedures, (LNF or TIF) and agree to have their standard GI medical data for 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness as measured by a 75% reduction in GERD HRQL) | 3 years
  To compare the effectiveness of TIF and LNF at the end of three years compared to baseline using a 75% reduction in GERD Health-related Quality of Life (GERD-HRQL) as a threshold for effectiveness.

SECONDARY OUTCOMES:
Effectiveness using a 50% reduction in GERD-HRQL | 3 years
  Compare effectiveness using a 50% reduction in GERD-HRQL as a threshold for effectiveness of TIF and LNF at the end of three years compared to baseline.

OTHER OUTCOMES:
Durability of GERD surgeries | 1 year and 3 years
  Compare the durability of TIF to LNF by determining the proportion of patients that achieve either a) >75% or b) >50% within the first year that maintain this effect at three years
Comparison of TIF to LNF for Patient reported symptoms | 3 years
  Compare TIF to LNF with respect to other reported GI symptoms, complications and side effects.
Comparison of Post-Procedure cost | 3 years
  Estimate the post-procedure costs associated with episodes of care and any ensuing complications or side effects of TIF and LNF.

CONTACTS AND LOCATIONS:
Overall Officials: M. Brian Fennerty, M.D., Principal Investigator — Oregon Health and Science University; W. Scott Melvin, M.D., Principal Investigator — Montefiore Medical Center; Ashish Atreja, M.D., Study Chair — MOUNT SINAI HOSPITAL
Locations (10):
- United States (10):
  - OC Reflux, Huntington Beach, California
  - SurgOne Foregut Institute, Englewood, Colorado
  - GI Solutions Inc, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Lenox Hill Hospital, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas at Houston, Bellaire, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Reston Hospital Center/ GW University, Reston, Virginia